CLINICAL TRIAL: NCT01369069
Title: Stroke Hyperglycemia Insulin Network Effort (SHINE) Trial
Acronym: SHINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Neurological Emergencies Treatment Trials Network (NETT) (Network); Medical University of South Carolina (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Karen C. Johnston, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15959; U01NS069498 (NIH)
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Acute Ischemic Stroke; Diabetes; Hyperglycemia
Keywords: stroke; diabetes; hyperglycemia
MeSH Terms: conditions — Ischemic Stroke; Diabetes Mellitus; Hyperglycemia; Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV insulin drip with target glucose 80 mg/dL - 130 mg/dL (Experimental): The intervention arm will have a targeted glucose concentration of 80-130 mg/dL. IV insulin drip will be titrated to keep glucose concentration in this range.
  Interventions: Drug: IV insulin to maintain target glucose concentration of 80-130 mg/dL
- Sub Q insulin to keep glucose less than 180 mg/dL (Active Comparator): This standard care arm will get sub q insulin sliding scale to keep glucose concentration less than 180 mg/dL
  Interventions: Drug: Standard Care control - sliding scale insulin to keep glucose less than 180 mg/dL

INTERVENTIONS:
Drug: IV insulin to maintain target glucose concentration of 80-130 mg/dL — Intervention is to keep glucose concentration 80-130 mg/dL for up to 72 hours after randomization. IV insulin drip will be used to maintain glucose target.
  Other Names: Continuous intravenous insulin
  Arms: IV insulin drip with target glucose 80 mg/dL - 130 mg/dL
Drug: Standard Care control - sliding scale insulin to keep glucose less than 180 mg/dL — Sliding scale sub q insulin given will be given up to 4 times per day based on glucose concentration. It will be given only if glucose concentration greater than or equal to 180 mg/dL.
  Other Names: Sliding scale insulin
  Arms: Sub Q insulin to keep glucose less than 180 mg/dL

SUMMARY:
The Stroke Hyperglycemia Insulin Network Effort (SHINE) Trial is a multicenter, randomized, controlled clinical trial of 1400 patients that will include approximately 60 enrolling sites. The study hypotheses are that treatment of hyperglycemic acute ischemic stroke patients with targeted glucose concentration (80mg/dL - 130 mg/dL) will be safe and result in improved 3 month outcome after stroke.

DETAILED DESCRIPTION:
Eligible subjects must be randomized within 12 hours of stroke symptom onset and either have type 2 diabetes and glucose concentrations of over 110 mg/dL or no history of diabetes and glucose concentrations of 150 mg/dL or higher on initial evaluation. The enrolling sites include the Neurological Emergencies Treatment Trials (NETT) sites as well as non NETT sites from all over the United States. The study evaluates the safety and efficacy of targeted glucose control (treatment group - IV insulin with target 80-130 mg/dl) verses control therapy of sub q insulin plus basal insulin with target glucose less than 180 mg/ dL.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Clinical diagnosis of ischemic stroke defined as acute neurological deficit occurring in one or more cerebral vascular territories. Neuroimaging must be done to exclude intracranial hemorrhage (ICH).
3. Randomization must be within 12 hours after stroke symptom onset and treatment is recommended, but not required, to begin within 3 hours after hospital arrival. If time of symptom onset is unclear or patient is awakening with stroke symptoms, the time of onset will be the time the patient was last known to be normal.
4. Known history of type 2 diabetes mellitus and glucose >110 mg/dL OR admission blood glucose ≥150 mg/dL in those w/o known diabetes mellitus
5. Baseline NIHSS score of 3-22
6. Pre-stroke modified Rankin Scale score = 0 for patients with an NIHSS score of 3-7. Pre-stroke modified Rankin Scale score = 0 or 1 for patients with an NIHSS score of 8-22.
7. Able to provide a valid informed consent to be in the study (self or their authorized legally accepted representative). The approved consent form must be signed and dated in accordance with federal and institutional guidelines.

Exclusion Criteria:

1. Known history of type 1 diabetes mellitus
2. Substantial pre-existing neurological or psychiatric illness that would confound the neurological assessment or other outcome assessment
3. Having received experimental therapy for the enrollment stroke. IV tPA (up to 4.5 hrs) or IA tPA are allowed as are IA therapies including use of FDA cleared devices. Non FDA cleared devices are considered experimental and are excluded.
4. Pregnant or breast-feeding at the time of study entry
5. Other serious conditions that make the patient unlikely to survive 90 days
6. Inability to follow the protocol or return for the 90 day follow up
7. Renal dialysis (including hemo or peritoneal dialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1151 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen C Johnston, MD, MSc, Study Chair — University of Virginia; Christiana Hall, MD, MS, Principal Investigator — UT Southwestern; Askiel Bruno, MD, MS, Principal Investigator — Augusta University; Valerie Durkalski, PhD, Principal Investigator — Medical University of South Carolina; William Barsan, MD, Principal Investigator — University of Michigan; Kevin Barrett, MD, Principal Investigator — Mayo Clinic
Locations (70):
- United States (70):
  - University of Arizona Medical Center - South Campus, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - Long Beach Memorial Medical Center, Long Beach, California
  - Ronald Regan Medical Center, Los Angeles, California
  - San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center - Davies Campus, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Emory University Hospital - Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital-Troy, Troy, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - JFK Medical Center, Edison, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Kings County Hospital, Brooklyn, New York
  - SUNY Downstate University Hospital of Brooklyn, Brooklyn, New York
  - Buffalo General Medical Center, Buffalo, New York
  - The Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Maimonides Medical Center, New York, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Summa Akron City Hospital, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Wexner Medical Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC - Mercy, Pittsburgh, Pennsylvania
  - WellSpan York Hospital, York, Pennsylvania
  - St. Thomas Neuroscience Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Seton Medical Center at UT, Austin, Texas
  - Seton Medical Center, Austin, Texas
  - UT Southwestern-Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern-Zale Lipshy University Hospital, Dallas, Texas
  - Valley Baptist Medical Center, Harlingen, Texas
  - Baylor College of Medicine, Houston, Texas
  - Memorial Herman Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Froedtert Memorial Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Result] Johnston KC, Bruno A, Pauls Q, Hall CE, Barrett KM, Barsan W, Fansler A, Van de Bruinhorst K, Janis S, Durkalski-Mauldin VL; Neurological Emergencies Treatment Trials Network and the SHINE Trial Investigators. Intensive vs Standard Treatment of Hyperglycemia and Functional Outcome in Patients With Acute Ischemic Stroke: The SHINE Randomized Clinical Trial. JAMA. 2019 Jul 23;322(4):326-335. doi: 10.1001/jama.2019.9346. PMID 31334795
- [Derived] Southerland AM, Mayer SA, Chiota-McCollum NA, Bolte AC, Pauls Q, Pettigrew LC, Bleck TP, Conaway M, Johnston KC. Glucose Control and Risk of Symptomatic Intracerebral Hemorrhage Following Thrombolysis for Acute Ischemic Stroke: A SHINE Trial Analysis. Neurology. 2024 May 14;102(9):e209323. doi: 10.1212/WNL.0000000000209323. Epub 2024 Apr 16. PMID 38626363
- [Derived] Arteaga DF, Ulep R, Kumar KK, Southerland AM, Conaway MR, Faber J, Wintermark M, Joyner D, Sharashidze V, Hirsch K, Giurgiutiu DV, Hannawi Y, Aziz Y, Shutter L, Visweswaran A, Williams A, Williams K, Gunter S, Haughey HM, Bruno A, Johnston KC, Patel VN; SHINE Trial Investigators. Collateral status, hyperglycemia, and functional outcome after acute ischemic stroke. BMC Neurol. 2022 Nov 4;22(1):408. doi: 10.1186/s12883-022-02943-4. PMID 36333676
- [Derived] Connor JT, Broglio KR, Durkalski V, Meurer WJ, Johnston KC. The Stroke Hyperglycemia Insulin Network Effort (SHINE) trial: an adaptive trial design case study. Trials. 2015 Mar 4;16:72. doi: 10.1186/s13063-015-0574-8. PMID 25885963
- [Derived] Garofolo KM, Yeatts SD, Ramakrishnan V, Jauch EC, Johnston KC, Durkalski VL. The effect of covariate adjustment for baseline severity in acute stroke clinical trials with responder analysis outcomes. Trials. 2013 Apr 11;14:98. doi: 10.1186/1745-6215-14-98. PMID 24499406
- [Derived] Bruno A, Durkalski VL, Hall CE, Juneja R, Barsan WG, Janis S, Meurer WJ, Fansler A, Johnston KC; SHINE investigators. The Stroke Hyperglycemia Insulin Network Effort (SHINE) trial protocol: a randomized, blinded, efficacy trial of standard vs. intensive hyperglycemia management in acute stroke. Int J Stroke. 2014 Feb;9(2):246-51. doi: 10.1111/ijs.12045. Epub 2013 Mar 19. PMID 23506245
- See also: General information of trial — https://nett.umich.edu/clinical-trials/shine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2012 and August 2018, a total of 70 United States sites were included in the trial, and 63 sites enrolled at least one patient.
Pre-assignment Details: 28977 patients were excluded after screening. Of those, 27344 did not meet eligibility criteria; 1156 were unable to provide informed consent or refused participation; 342 had other reasons and 135 did not specify a reason.
Period: Overall Study
Arm/Group | IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL | Sub Q Insulin to Keep Glucose Less Than 180 mg/dL
Started | 581 | 570
Completed | 564 | 554
Not Completed | 17 | 16
Not completed — Lost to Follow-up | 8 | 9
Not completed — Withdrawal by Subject | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL | Sub Q Insulin to Keep Glucose Less Than 180 mg/dL | Total
Number analyzed (Participants) | 581 | 570 | 1151
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [57 to 75] | 66 [57 to 76] | 66 [57 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 260 | 264 | 524
  Male | 321 | 306 | 627
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 87 | 91 | 178
  Not Hispanic or Latino | 460 | 449 | 909
  Unknown or Not Reported | 34 | 30 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 12 | 18 | 30
  Native Hawaiian or Other Pacific Islander | 2 | 5 | 7
  Black or African American | 180 | 154 | 334
  White | 366 | 368 | 734
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 23 | 44
Final diagnosis [Count of Participants; unit: Participants]
  Ischemic stroke | 542 | 524 | 1066
  Transient ischemic attack | 8 | 12 | 20
  Other | 31 | 34 | 65
Thrombolysis or Thrombectomy [Count of Participants; unit: Participants]
  Intravenous tPA | 372 | 353 | 725
  Mechanical treatment | 74 | 72 | 146
  Intraarterial drug therapy | 14 | 21 | 35
  None | 121 | 124 | 245
Medical History [Count of Participants; unit: Participants]
  Hypertension | 513 | 502 | 1015
  Diabetes mellitus (Type 2) | 468 | 455 | 923
  Hyperlipidemia | 350 | 327 | 677
  Coronary artery disease | 159 | 167 | 326
  Atrial fibrillation | 124 | 106 | 230
  Previous Ischemic stroke | 104 | 99 | 203
  Previous large vessel atherosclerosis | 42 | 39 | 81
Eligibility POC blood glucose (mg/dL) [Median (Inter-Quartile Range); unit: mg/dL] | 188 [153 to 250] | 187 [155 to 248] | 187.5 [154 to 250]
Baseline NIHSS at randomization [Median (Inter-Quartile Range); unit: NIHSS score range: 0 to 42] | 7 [5 to 12] | 7 [5 to 13] | 7 [5 to 13]
Baseline NIHSS category at randomization [Count of Participants; unit: Participants]
  Mild (NIHSS 3-7) | 291 | 291 | 582
  Moderate (NIHSS 8-14) | 177 | 158 | 335
  Severe (NIHSS 15-22) | 113 | 121 | 234

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Favorable Modified Rankin Scale (Yes/No)
Description: Favorable for the primary efficacy outcome is defined as modified Rankin Scale (mRS) score of 0 in patients with mild stroke (baseline NIHSS 3-7), mRS 0 or 1 in patients with moderate stroke (baseline NIHSS 8-14), and mRS 0, 1 or 2 in patients with severe stroke (baseline NIHSS 15-22) at 90 days with a pre-specified range of acceptable days of 76 -120 days. The mRS is a stroke outcome scale used to assess functional status after stroke. It consists of seven levels (0-6) where 0 indicates no residual symptoms at all, 5 indicates severe disability and 6 indicates death. The person collecting the mRS score was to be blinded to the participant's treatment group assignment.
Time Frame: 90 days (-14/+30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL | Sub Q Insulin to Keep Glucose Less Than 180 mg/dL
Number analyzed (Participants) | 581 | 570
Participants | 119 | 123
Statistical Analysis 1: Comparison: IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL vs Sub Q Insulin to Keep Glucose Less Than 180 mg/dL; It was hypothesized that intensive blood glucose control would be efficacious and safe in acute ischemic stroke patients compared to standard glucose control; Test type: Superiority; p = 0.55, Regression, Logistic — The a priori threshold for statistical significance was 0.05; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.87 to 1.08] — Adjusted for baseline NIHSS strata (3-7, 8-14, 15-22) and thrombolysis use (Yes/No; includes both IV and IA therapies). Multiple imputation was used for missing data

2. Primary Outcome: Number of Participants With Severe Hypoglycemia (Blood Glucose < 40mg/dL)
Description: Severe hypoglycemia (blood glucose < 40mg/dL) is the primary safety outcome and will be measured during the 72 hour treatment period.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL | Sub Q Insulin to Keep Glucose Less Than 180 mg/dL
Number analyzed (Participants) | 581 | 570
Participants | 15 | 0
Statistical Analysis 1: Comparison: IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL vs Sub Q Insulin to Keep Glucose Less Than 180 mg/dL; Test type: Superiority; p < 0.001, Fisher Exact; Risk Difference (RD) = 2.58, 95% CI 2-sided [1.29 to 3.87] — The data of the estimation parameter and the confidence intervals were presented as percentages

3. Secondary Outcome: Number of Participants With a Favorable NIHSS
Description: The NIHSS (National Institutes of Health Stroke Scale) score ranges from 0 to 42, with higher scores indicating greater neurological deficits. A favorable NIHSS was defined as a score of 0 or 1 on the NIHSS at 90 days post randomization.
Time Frame: Follow up (Max 164 days)
Measure: Count of Participants; unit: Participants
Arm/Group | IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL | Sub Q Insulin to Keep Glucose Less Than 180 mg/dL
Number analyzed (Participants) | 348 | 371
Participants | 152 | 166
Statistical Analysis 1: Comparison: IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL vs Sub Q Insulin to Keep Glucose Less Than 180 mg/dL; Test type: Superiority; p = 0.77, Chi-squared; Risk Difference (RD) = -1.07, 95% CI 2-sided [-8.33 to 6.20] — The data of the estimation parameter and the confidence intervals were presented as percentages

4. Secondary Outcome: Number of Participants With a Favorable Barthel Index
Description: Favorable outcomes for the Barthel Index was defined as a score of 95-100 on the BI at 90 days post randomization. Barthel - Barthel Index for Activities of Daily Living (ADL) assesses functional independence, generally in stroke patients. Scores range from 0-100 with higher scores indicating greater ability to perform activities of daily living.
Time Frame: Follow up (Max 164 days)
Measure: Count of Participants; unit: Participants
Arm/Group | IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL | Sub Q Insulin to Keep Glucose Less Than 180 mg/dL
Number analyzed (Participants) | 491 | 477
Participants | 271 | 261
Statistical Analysis 1: Comparison: IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL vs Sub Q Insulin to Keep Glucose Less Than 180 mg/dL; Test type: Superiority; p = 0.88, Chi-squared; Risk Difference (RD) = 0.48, 95% CI 2-sided [-5.79 to 6.75] — The data of the estimation parameter and the confidence intervals were presented as percentages

5. Secondary Outcome: Stroke Specific Quality of Life (SSQOL)
Description: Stroke Specific Quality of Life. Scores range from 1-5 with higher scores indicating better quality of life
Time Frame: Follow up (Max 164 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL | Sub Q Insulin to Keep Glucose Less Than 180 mg/dL
Number analyzed (Participants) | 442 | 432
score on a scale | 3.75 [2.98 to 4.40] | 3.69 [3.02 to 4.46]
Statistical Analysis 1: Comparison: IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL vs Sub Q Insulin to Keep Glucose Less Than 180 mg/dL; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.06, 95% CI 2-sided [-0.13 to 0.25]

6. Other Pre Specified Outcome: Death
Description: Death from any cause
Time Frame: 90 days (+30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL | Sub Q Insulin to Keep Glucose Less Than 180 mg/dL
Number analyzed (Participants) | 581 | 570
Participants | 54 | 65
Statistical Analysis 1: Comparison: IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL vs Sub Q Insulin to Keep Glucose Less Than 180 mg/dL; Test type: Superiority; p = 0.24, Chi-squared; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.58 to 1.15]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were assessed and reported through the treatment period (up to 72 hours). Serious adverse events were reported throughout the study period (randomization through end of study; end of study was 90 days post randomization or earlier if a participant died or withdrew consent).
Arm/Group | IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL | Sub Q Insulin to Keep Glucose Less Than 180 mg/dL
All-Cause Mortality (participants affected / at risk) | 54/581 | 65/570
Serious Adverse Events (participants affected / at risk) | 209/581 | 198/570
Other Adverse Events (participants affected / at risk) | 384/581 | 134/570
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL (N=581) | Sub Q Insulin to Keep Glucose Less Than 180 mg/dL (N=570)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Other (combined AEs happened only once) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 6 (6) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 8 (9) | 4 (4)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 7 (10) | 7 (7)
Cardiac failure (Cardiac disorders) | 3 (4) | 5 (5)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 6 (6) | 5 (5)
Other (combined AEs happened only once) (Cardiac disorders) | 1 (1) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (2) | 3 (3)
Other (combined AEs happened only once) (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Other (combined AEs happened only once) (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other (combined AEs happened only once) (Gastrointestinal disorders) | 2 (2) | 6 (6)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 2 (2) | 3 (4)
Device occlusion (General disorders) | 0 (0) | 2 (2)
Multi-organ failure (General disorders) | 2 (2) | 1 (1)
Other (combined AEs happened only once) (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (2) | 3 (3)
Sudden death (General disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Other (combined AEs happened only once) (Hepatobiliary disorders) | 2 (2) | 1 (1)
Other (combined AEs happened only once) (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Other (combined AEs happened only once) (Infections and infestations) | 5 (5) | 3 (3)
Pneumonia (Infections and infestations) | 15 (16) | 14 (14)
Sepsis (Infections and infestations) | 7 (7) | 14 (15)
Septic shock (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (7) | 4 (4)
Urosepsis (Infections and infestations) | 1 (1) | 2 (2)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Other (combined AEs happened only once) (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 7 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 21 (28) | 2 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Other (combined AEs happened only once) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Other (combined AEs happened only once) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Other (combined AEs happened only once) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Brain oedema (Nervous system disorders) | 10 (10) | 11 (11)
Cerebral haemorrhage (Nervous system disorders) | 4 (5) | 4 (4)
Cerebrovascular accident (Nervous system disorders) | 10 (10) | 12 (12)
Convulsion (Nervous system disorders) | 7 (7) | 8 (8)
Embolic stroke (Nervous system disorders) | 3 (3) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 4 (5)
Haemorrhage intracranial (Nervous system disorders) | 4 (4) | 4 (4)
Haemorrhagic transformation stroke (Nervous system disorders) | 36 (37) | 27 (28)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 16 (16) | 16 (21)
Neurological decompensation (Nervous system disorders) | 7 (7) | 17 (18)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Other (combined AEs happened only once) (Nervous system disorders) | 3 (3) | 2 (2)
Stroke in evolution (Nervous system disorders) | 9 (9) | 11 (11)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 4 (5) | 4 (4)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 2 (3) | 0 (0)
Other (combined AEs happened only once) (Psychiatric disorders) | 1 (1) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (3)
Other (combined AEs happened only once) (Renal and urinary disorders) | 1 (1) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 8 (8) | 7 (7)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other (combined AEs happened only once) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (8)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 10 (10)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Other (combined AEs happened only once) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 1 (1)
Other (combined AEs happened only once) (Surgical and medical procedures) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 4 (5) | 3 (3)
Embolism (Vascular disorders) | 2 (2) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 5 (5) | 2 (2)
Other (combined AEs happened only once) (Vascular disorders) | 2 (2) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Insulin Drip With Target Glucose 80 mg/dL - 130 mg/dL (N=581) | Sub Q Insulin to Keep Glucose Less Than 180 mg/dL (N=570)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 9 (9) | 9 (9)
Bradycardia (Cardiac disorders) | 3 (3) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Other (combined AEs happened only once) (Cardiac disorders) | 2 (2) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Other (combined AEs happened only once) (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Other (combined AEs happened only once) (Eye disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Other (combined AEs happened only once) (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (6) | 8 (8)
Catheter site haematoma (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2)
Other (combined AEs happened only once) (General disorders) | 3 (3) | 2 (2)
Pain (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 7 (7) | 5 (5)
Other (combined AEs happened only once) (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Other (combined AEs happened only once) (Infections and infestations) | 1 (1) | 4 (4)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 12 (12) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Other (combined AEs happened only once) (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1)
Blood chloride increased (Investigations) | 3 (3) | 2 (2)
Blood cholesterol increased (Investigations) | 2 (2) | 1 (1)
Blood creatinine decreased (Investigations) | 1 (1) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 1 (1)
Carbon dioxide decreased (Investigations) | 2 (2) | 0 (0)
High density lipoprotein decreased (Investigations) | 2 (2) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Other (combined AEs happened only once) (Investigations) | 8 (12) | 9 (12)
Red cell distribution width increased (Investigations) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 3 (3) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 311 (574) | 16 (26)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (14) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Other (combined AEs happened only once) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other (combined AEs happened only once) (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Brain oedema (Nervous system disorders) | 5 (5) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 2 (2)
Haemorrhagic transformation stroke (Nervous system disorders) | 23 (23) | 13 (13)
Headache (Nervous system disorders) | 11 (12) | 7 (7)
Neurological decompensation (Nervous system disorders) | 10 (11) | 8 (8)
Neurological symptom (Nervous system disorders) | 2 (2) | 0 (0)
Other (combined AEs happened only once) (Nervous system disorders) | 6 (6) | 2 (2)
Stroke in evolution (Nervous system disorders) | 2 (2) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Other (combined AEs happened only once) (Psychiatric disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Other (combined AEs happened only once) (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 4 (4) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Other (combined AEs happened only once) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Other (combined AEs happened only once) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 4 (4) | 5 (5)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)
Hypotension (Vascular disorders) | 5 (5) | 4 (4)
Malignant hypertension (Vascular disorders) | 1 (1) | 1 (1)
Other (combined AEs happened only once) (Vascular disorders) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-10-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT01369069/Prot_000.pdf
  • Statistical Analysis Plan (2015-01-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT01369069/SAP_001.pdf